CLINICAL TRIAL: NCT05628389
Title: Phone Enabled Implementation of Cessation Support
Acronym: PHOENICS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB202202537 -N; R01CA262319 (NIH)
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ask-Advice-Assist (AAA) (Other): All patients will be screened for tobacco use, and offer brief cessation advice and counseling.
  Interventions: Behavioral: Educational materials; Behavioral: Provider training; Behavioral: Electronic reminders
- Ask-Advise-Connect (AAC) (Experimental): Patients in will be connected to phone counseling and will receive six sessions of telephone counseling.
  Interventions: Behavioral: Educational materials; Behavioral: Phone counseling; Behavioral: Provider training; Behavioral: Electronic reminders
- Ask-Advise-Connect (AAC) + Nicotine Replacement Therapy (NRT) (Experimental): In addition to AAC, patients will be offered NRT.
  Interventions: Behavioral: Educational materials; Behavioral: Phone counseling; Drug: Nicotine Replacement Therapy; Behavioral: Provider training; Behavioral: Electronic reminders

INTERVENTIONS:
Behavioral: Educational materials — Patient educational materials to address insufficient knowledge about harms of tobacco use and cessation.
Behavioral: Phone counseling — Cessation counseling to address insufficient patient self-efficacy and motivation.
  Arms: Ask-Advise-Connect (AAC); Ask-Advise-Connect (AAC) + Nicotine Replacement Therapy (NRT)
Drug: Nicotine Replacement Therapy — Nicotine patches to address nicotine withdrawal symptoms in patients.
  Arms: Ask-Advise-Connect (AAC) + Nicotine Replacement Therapy (NRT)
Behavioral: Provider training — Provider training to address insufficient knowledge and self-efficacy to deliver AAA/AAC to patients.
Behavioral: Electronic reminders — Electronic reminders to address the lack of integration of AAA/AAC into practice.

SUMMARY:
The tobacco use burden in Lebanon is exceptionally high: 35% of adults are current cigarette smokers and 39% are current waterpipe smokers. Although the World Health Organization endorses evidence-based interventions for population-level tobacco dependence treatment, recommended treatments are not integrated as a routine part of primary care in Lebanon, as is the case in other low-resource settings. The objective of this proposal is to evaluate the comparative effectiveness of promising multi-component interventions for implementing evidence-based cessation treatment in Lebanon's national system of primary health care centers.

DETAILED DESCRIPTION:
The research team will conduct a group-randomized trial comparing three arms: 1) Ask about tobacco use, advise to quit, assist with brief counseling (AAA) as standard care; 2) Ask, advise, connect to phone-based counseling (AAC); and 3) AAC+ Nicotine Replacement Therapy (NRT). Our central hypothesis is that connecting patients to phone-based counseling with cessation medication is the most effective alternative. The hybrid design is informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework which emphasizes key steps and multilevel factors to optimize implementation success. The following specific aims will be pursued: 1) adapt and tailor an existing smoking cessation program to deliver phone-based counseling to smokers in Lebanon; 2) test the effectiveness and cost-effectiveness of a referral-based program that delivers smoking cessation services to primary care patients; and 3) identify the multilevel determinants of implementation and sustainability using mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* A current daily cigarette smoker and/or a regular waterpipe smoker (smokes at least 1-2 times/week).
* Not pregnant
* Reachable by phone
* Interested in quitting
* Lives in Greater Beirut Area

Exclusion Criteria:

* Patients who use other tobacco products including vape exclusively.
* Any patient below 18 years old.
* Cigarette smokers who do not smoke on daily basis.
* Waterpipe smokers who smoke less than once/weekly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
7-day smoking abstinence | 6 Months
  Carbon monoxide confirmed-abstinence from smoking in the last 7 days days prior to assessment

OTHER OUTCOMES:
Self-reported abstinence | 1, 3, 6 months
  Continuous abstinence, quit attempts, smoking reduction

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Salloum, PhD, Principal Investigator — University of Florida
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salloum RG, Romani M, Bteddini DS, El-Jardali F, Lee JH, Theis R, LeLaurin JH, Hamadeh R, Osman M, Abla R, Khaywa J, Ward KD, Shelley D, Nakkash R. An effectiveness-implementation hybrid trial of phone-based tobacco cessation interventions in the Lebanese primary healthcare system: protocol for project PHOENICS. Implement Sci Commun. 2023 Jun 26;4(1):72. doi: 10.1186/s43058-023-00456-w. PMID 37365656